CLINICAL TRIAL: NCT01282021
Title: Molecular Immunohematology in Ethiopian Sub-Populations
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999911086; 11-CC-N086
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Immunohematology
Keywords: Serologic RBC Antigens; RBC Antigen Molecular Studies; Blood Transfusion; RBC Antigen Profiles; Alloimmunization; Natural History

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Region 1: Northern part: Gonder, Gojam, Tigray
- Region 2: Southern Ethiopia: Bale, Sidamo, Gambela
- Region 3: Northeastern and Southeastern Ethiopia

SUMMARY:
Alloimmunization to blood products in transfused patients is a recognized management challenge in the clinical setting. In particular the ethnic and racial specificity of RBC antigens and the limited availability of matched healthy volunteer blood donors have intensified the dilemma. The presence of low prevalence clinically significant RBC antigens among minorities account for the higher rate of alloimmunization observed in patients from this group. This is partly due to the racial and ethnic differences between the blood donor and recipient populations in the U.S.

The increasing number of new Ethiopian-American immigrants in the US presenting to the health care system with blood transfusion requirements makes understanding the unique transfusion needs of this minority population imperative. Although the majority of African Americans claim origin to West Africa, Ethiopians, being from East Africa, represent a rapidly growing population in the United States. Furthermore, identifying genetic similarities and disparities to their West African counterparts will certainly have clinical implications in terms of transfusion support and disease modifiers. This additional information would help in understanding the natural history and transfusion requirements of certain debilitating diseases, such as Sickle Cell Disease (SCD), which are known to occur more commonly in African Americans. Identifying ethnically and racially similar individuals could assist in recruiting healthy volunteer donors with similar RBC antigen profiles potentially supplementing the rare donor pool.

Although extensive archeological and sporadic serologic RBC antigen studies have been conducted in Ethiopia, there are no population wide RBC antigen molecular studies. Our study population is selected by altitude and migration history. Ethiopia, being in close proximity to the Red Sea in the northeast, Indian Ocean in the southeast and the rest of Africa in the south/west has diverse population.

The study is a population based analysis of genetic variation of blood group antigens in three distinct and conserved Ethiopian sub-populations. Statistical analysis using Chi-square tests will be performed for each blood group antigen to detect differences in the distribution between the three sub-populations. The The Lead Associate Investigator (LAI), and, as appropriate, additional Investigators, will travel to Ethiopia to collect blood samples, which will be analyzed in the Department of Transfusion Medicine (DTM) at the National Institutes of Health (NIH) using the standard serologic methods and currently available molecular genotyping systems. Samples will also be stored for future high throughput sequencing analysis and other studies.

The study will be a systematic analysis of the distribution of blood group antigens in Ethiopian sub-populations. Furthermore, new variants could be detected allowing insight into the correlation of particular genotypes and phenotypes.

DETAILED DESCRIPTION:
Alloimmunization to blood products in transfused patients is a recognized management challenge in the clinical setting. In particular the ethnic and racial specificity of RBC antigens and the limited availability of matched healthy volunteer blood donors have intensified the dilemma. The presence of low prevalence clinically significant RBC antigens among minorities account for the higher rate of alloimmunization observed in patients from this group. This is partly due to the racial and ethnic differences between the blood donor and recipient populations in the U.S.

The increasing number of new Ethiopian-American immigrants in the US presenting to the health care system with blood transfusion requirements makes understanding the unique transfusion needs of this minority population imperative. Although the majority of African Americans claim origin to West Africa, Ethiopians, being from East Africa, represent a rapidly growing population in the United States. Furthermore, identifying genetic similarities and disparities to their West African counterparts will certainly have clinical implications in terms of transfusion support and disease modifiers. This additional information would help in understanding the natural history and transfusion requirements of certain debilitating diseases, such as Sickle Cell Disease (SCD), which are known to occur more commonly in African Americans. Identifying ethnically and racially similar individuals could assist in recruiting healthy volunteer donors with similar RBC antigen profiles potentially supplementing the rare donor pool.

Although extensive archeological and sporadic serologic RBC antigen studies have been conducted in Ethiopia, there are no population wide RBC antigen molecular studies. Our study population is selected by altitude and migration history. Ethiopia, being in close proximity to the Red Sea in the northeast, Indian Ocean in the southeast and the rest of Africa in the south/west has diverse population.

The study is a population based analysis of genetic variation of blood group antigens in three distinct and conserved Ethiopian sub-populations. Statistical analysis using Chi-square tests will be performed for each blood group antigen to detect differences in the distribution between the three sub-populations. The The Lead Associate Investigator (LAI), and, as appropriate, additional Investigators, will travel to Ethiopia to collect blood samples, which will be analyzed in the Department of Transfusion Medicine (DTM) at the National Institutes of Health (NIH) using the standard serologic methods and currently available molecular genotyping systems. Samples will also be stored for future high throughput sequencing analysis and other studies.

The study will be a systematic analysis of the distribution of blood group antigens in Ethiopian sub-populations. Furthermore, new variants could be detected allowing insight into the correlation of particular genotypes and phenotypes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers >= 18 year of age. Volunteer healthy donors above the age of 18 years, who have lived in the area since birth, and are at least 6 or 7 generation from endogenous families in the region, will be recruited. A detailed ancestral line of descent (pedigree) is not mandatory to the study and will not be performed. Individuals residing in rural regions are mostly conserved and it may be possible that some donors could be closely related. However, to identify as diverse a population of potential blood donors as possible, and avoid dilution of ancestral genes blood samples will be collected from individuals known to reside in the region for generations and not known to be closely related. Donors will be recruited through the local schools, churches, and community organizations. The oral consent will include a question where each donor will be asked if anyone in his/her family is also donating a sample, and, if so, how close the relationship is to that individual. Blood collection will be on a firstcome, first serve basis; individuals will be made aware that only one person among a group of close relatives will be included in the study.

EXCLUSION CRITERIA:

Individuals < 18 years of age will be excluded from the study. The study is a population study and the information obtained from individuals above 18 years is not expected to be different from those who are under 18 years old. Also, the need to involve adults to consent individuals under 18 years old would be complicated. All donors should be healthy volunteer individuals at the time of sample collection. Any potential donor with physical and mental disability, individuals with known infectious and/or non-infectious diseases, and pregnant women, are excluded from the study.

The study will be conducted in coordination with Addis Ababa University Medical Faculty and the regional Health Offices in collaboration with Ethiopian Red Cross. The local PI, Dr. Amha Gebgremedhin, is a member of the Addis Ababa University Medical faculty, Department of Hematology, residing in Addis Ababa. The local health centers in the three regions listed above will be used as centers for sample collection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of three distinct and conserved Ethiopian sub-populations.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2012-11-03 (Actual)

PRIMARY OUTCOMES:
Serum Collection | 10 years
  To elucidate the molecular distribution of blood group alleles predicting RBC antigens in three different sub-populations in Ethiopia.

CONTACTS AND LOCATIONS:
Overall Officials: Willy A Flegel, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- Addis Ababa University, Addis Ababa, Ethiopia

REFERENCES:
- [Background] Daly MG, Frampton CM, Troughton RW. Improving risk stratification for heart failure. A role for serial testing of B-type natriuretic peptides? J Am Coll Cardiol. 2010 Feb 2;55(5):451-3. doi: 10.1016/j.jacc.2009.08.060. No abstract available. PMID 20117458
- [Background] Rademakers FE, Bogaert J. Cardiac dysfunction in heart failure with normal ejection fraction: MRI measurements. Prog Cardiovasc Dis. 2006 Nov-Dec;49(3):215-27. doi: 10.1016/j.pcad.2006.08.012. PMID 17084181
- [Background] Mann DL. Mechanisms and models in heart failure: A combinatorial approach. Circulation. 1999 Aug 31;100(9):999-1008. doi: 10.1161/01.cir.100.9.999. No abstract available. PMID 10468532
- [Derived] Srivastava K, Yin Q, Makuria AT, Rios M, Gebremedhin A, Flegel WA. CD59 gene: 143 haplotypes of 22,718 nucleotides length by computational phasing in 113 individuals from different ethnicities. Transfusion. 2024 Jul;64(7):1296-1305. doi: 10.1111/trf.17869. Epub 2024 May 30. PMID 38817044
- [Derived] Yin Q, Srivastava K, Schneider JB, Gebremedhin A, Makuria AT, Flegel WA. Molecular analysis of the ICAM4 gene in an autochthonous East African population. Transfusion. 2019 May;59(5):1880-1881. doi: 10.1111/trf.15217. Epub 2019 Feb 20. No abstract available. PMID 30790296